CLINICAL TRIAL: NCT06010589
Title: Bioequivalence Study to Compare the Pharmacokinetics and Safety Following Administration of DWJ1558 and Co-administration of DWC202310 and DWC202311 in Healthy Volunteers
Brief Title: Bioequivalence Study for the Safety and the Pharmacokinetics of DWJ1558 in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1558101
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: DWJ1558 (Experimental)
  Interventions: Drug: DWJ1558
- Intervention: DWC202310 and DWC202311 (Experimental)
  Interventions: Drug: DWC202310 and DWC202311

INTERVENTIONS:
Drug: DWJ1558 — DWJ1558
  Arms: Intervention: DWJ1558
Drug: DWC202310 and DWC202311 — Co-administration of DWC202310 and DWC202311
  Arms: Intervention: DWC202310 and DWC202311

SUMMARY:
This study aims to compare the pharmacokinetics and safety following administration of DWJ1558 and co-administration of DWC202310 and DWC202311 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* over 19 year old

Exclusion Criteria:

* Pancreatitis
* Diabetic ketoacidosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss of DWJ1558 | At pre-dose (0 hour), and post-dose 1 to 72 hour.
  Maximum plasma concentration at steady-state(Cmax,ss) of DWJ1558
AUCt of DWJ1558 | At pre-dose (0 hour), and post-dose 1 to 72 hour.
  Area under the curve from the time of dosing to the last measurable concentration(AUCt) of DWJ1558

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus YANGJI Hospital, Seoul, South Korea